CLINICAL TRIAL: NCT06638385
Title: A Space-expanding Shield in Decompressive Hemicraniectomy for Stroke - a Randomized-controlled Multicenter Phase III Trial
Brief Title: A Space-expanding Shield in Decompressive Hemicraniectomy for Stroke
Acronym: SPACE SHIELD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPACE SHIELD
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: stroke; bone flap; cranioplasty
MeSH Terms: conditions — Stroke | interventions — delta 24-sterol reductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCE + SPACE SHIELD (Experimental): Patients in the experimental group receive a DCE with implantation of a space-expanding shield.
  Interventions: Procedure: DCE + SPACE SHIELD
- DCE + CP (Active Comparator): Patients in the control group receive a DCE similar to the intervention group, but without implantation of a space-expanding shield. Cranioplasty (CP) is performed after ~ 90 days in the customary manner.
  Interventions: Procedure: DCE + CP

INTERVENTIONS:
Procedure: DCE + SPACE SHIELD — Patients receive a DCE with implantation of a space-expanding shield.
  Arms: DCE + SPACE SHIELD
Procedure: DCE + CP — Patients in the control group receive a DCE similar to the intervention group, but without implantation of a space-expanding shield. Cranioplasty (CP) is performed after ~ 90 days in the customary manner.
  Arms: DCE + CP

SUMMARY:
Instead of the standard decompressive hemicraniectomy with subsequent cranioplasty a single surgery with the implantation of an individually molded space-expanding shield is investigated in for patients with increased intracranial pressure due to a malignant stroke.

DETAILED DESCRIPTION:
Background:

A malignant cerebral infarction causes edema resulting in a threatening increase of the intracranial pressure (ICP). Standard of care is a surgical removal of a part of the skull above the ischemic brain, the so-called decompressive hemicraniectomy (DCE). DCE allows the brain to swell, after detumescence of the brain parenchyma (usually several months later) the patients undergo a second surgery with implantation of either their own preserved bone flap or a bone flap substitute (a procedure referred to as cranioplasty (CP)).

Objective:

Despite its proven life-saving benefits, the strategy of DCE followed by CP carries several risks, among others

* Exposure of the brain parenchyma
* Various neurological deficits subsumed under the syndrome of the trephined
* Bone resorption: As shown in a previous prospective cohort study the above-mentioned risks may be prevented using an intraoperatively molded space-expanding protective shield, which is implanted and fixed directly after having performed (a so far customary) DCE. This shield allows the brain to swell while still providing protection.

SPACE SHIELD investigates whether the single-stage strategy of implanting a space-expanding shield represents a viable alternative to the standard DCE followed by CP."

Methods:

The inclusion of patients is planned to take place from January 2025 to December 2029. The study duration for the individual patients is 6 months. While the intervention group will be treated with the above-described space-expanding shield the control group will be treated with the customary DCE and following CP. The CP will be performed either with the original bone flap stored in customary manner or with a PMME bone flap. Examinations of the patients are planned after 1 - 7 days, 6 weeks, 3 months and 6 months after the initial surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant infarction of the middle cerebral artery identified by MRI including diffusion-weighted imaging or CT including perfusion imaging - fulfilling the European guidelines for decompressive hemicraniectomy (DCE) for stroke
* ≥ 18 and < 70 years of age
* Availability of consent from a next of kin and from the patient represented by an independent physician

Exclusion Criteria:

* Hyperacute need for DCE due to rapid neurological decline
* Contraindications to the use of polymethyl-methacrylate (PMMA), e.g., known hypersensitivity, allergy
* Known gentamicin allergy
* Pregnancy and active breast-feeding
* Patients with a former history of DCE and/or CP
* Active pulmonary or cranial infection
* Known coagulopathy independent of medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
modified Ranking Scale (mRS) score at 6 months | 6 months after surgery
  The primary outcome will be assessed by a blinded, independent, local study nurse.
  The sole task of this study nurse will be to assess the mRS based on a short interview with the patient.

SECONDARY OUTCOMES:
Number of further surgical interventions for ICP control | 6 months after surgery
  This includes surgical removal and exchange of the space-expanding shield, implantation of an EVD), surgery for further bony decompression, surgery for removal of hemorrhages or hygroma.
Occurrence of Hydrocephalus | 6 months after surgery
  Any radiological diagnosis of hydrocephalus requiring either a shunting procedure or an EVD, including revision, at least 2 weeks after study inclusion.
  Procedures before 2 weeks will qualify as an intervention for ICP control (a. Further surgical interventions for ICP control)
Number of Infections | 6 months after surgery
  Any infection leading to surgical revision and identification of bacteria by bacterial growth in microbacterial analysis from surgically obtained specimen. Wound healing difficulties treated with local treatment only (no surgical revision) will not count as infections.
Wound healing difficulties | 6 months after surgery
  Any surgery under general anaesthesia for wound healing difficulties, unless qualified as infection. The total number of events will be reported as well as the rate of patients with at least one event.
Syndrome of the trephined | 6 months after surgery
  The syndrome of the trephined subsumes various new or worsened neurological deficits attributed to the trephined state: headache, dizziness, fatigue, cognitive decline, decreased consciousness, sensory deficits, motor deficits, speech difficulties. It will be reported on the rate of patients experiencing the syndrome of the trephined, as well as to whether the patient's symptoms recovered following bone-flap re-insertion (fully, partially or not).
Overall survival at 6 months | 6 months after surgery
Cosmetic satisfaction at 6 months | 6 months after surgery
  The patient will be asked to self-evaluate the overall cosmetic results of the scar, shape of head and visible craniotomy edge using a 5-points Likert scale (very poor - poor - average - good - very good)
Quality of life score: EQ-5D-5L | 6 months after surgery
  EuroQoL 5D-5L questionnaire (Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/ Depression (rating from no problems to extreme problems) and health status self rating by patient (Score 0-100, 0 the worst health and 100 the best health))

CONTACTS AND LOCATIONS:
Overall Officials: Schucht Philippe, MD, Principal Investigator — Inselspital Bern, Department of Neurosurgery
Locations (6):
- Switzerland (6):
  - Kantonsspital Aarau, Aarau
  - Universitätsspital Basel, Basel
  - Inselspital Bern, Department of Neurosurgery, Bern
  - Luzerner Kantonsspital, Lucerne
  - Ente Ospedaliero Cantonale, Lugano
  - Kantonsspital St.Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No